CLINICAL TRIAL: NCT03020680
Title: The Effect of Redox Status on Bioavailability of Ubiquinone and Ubiquinol in 10 Older Adults
Brief Title: Bioavailability of Ubiquinone and Ubiquinol in Older Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Oliver Chen, Scientist I, Tufts University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2895
Record Dates: First submitted 2016-08-30; First posted 2017-01-13 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Absorption
MeSH Terms: interventions — coenzyme Q10

STUDY DESIGN:
Intervention Model Description: two 14-day intervention phases with a 2-week washout between each phase. randomized to receive 200mg/day ubiquinol or 200mg/day ubiquinone
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ubiquinol (Experimental): It is the reduced form of coenzyme Q10
  Interventions: Dietary Supplement: Coenzyme Q10
- ubiquinone (Active Comparator): It is the oxidized form of coenzyme Q10
  Interventions: Dietary Supplement: Coenzyme Q10

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 — To examine whether 200 mg/d ubiquinol for 14 days increase coenzyme Q10 status by a larger degree than 200 mg/d ubiquinone

SUMMARY:
Coenzyme Q10 (or CoQ10) is a marketed supplement in US even though it can be synthesized in the body via complicated biochemical pathways. It exists in both reduced and oxidized states, namely ubiquinol and ubiquinone, respectively. It is commonly present in all cell membranes. The main function of CoQ10 is to participate in energy production. Further, the reduced form of CoQ10, ubiquinol, is appreciated as an important lipophilic antioxidant to protect free radical induced damages to DNA, lipid, and proteins. Given that older adults have increased production of free radicals, suboptimal antioxidant defenses toward free radicals, and a decreased capability to replenish utilized CoQ10, CoQ10 supplementation can be one of feasible ways to increase CoQ10 status in order adults. Most supplements available for consumers are in the oxidized form. While the ubiquinol form is also available, whether the reduced form will be more effective to replenish CoQ10 status in older subjects remains to be explored. Thus, investigators aimed to examine whether ubiquinol will be more effectively absorbed in older adults with a low antioxidant defense status. To pursue this aim, investigators will conduct a double blind, randomized, crossover design trail with 5 study visits (1 screening visit and 4 study visits). Ten older men (>55 y, BMI: 25-5 kg/m2) with a compromised antioxidant defenses will be recruited and complete the trial. Eligible subjects will be randomized to receive 200 mg/d ubiquinol or ubiquinone for 2 weeks with 2-week washout between crossover. Ubiquinol and ubiquinone in plasma and immune cells in blood will be assessed to reveal whether the reduced form, ubiquinol, is more absorbable than the oxidized form, ubiquinone in older adults.

DETAILED DESCRIPTION:
Coenzyme Q10 (or CoQ10) is a marketed supplement in US even though it can be synthesized in the body via complicated biochemical pathways. It exists in both reduced and oxidized states, namely ubiquinol and ubiquinone, respectively. It is commonly present in all cell membranes. The main function of CoQ10 is to participate in energy production. Further, the reduced form of CoQ10, ubiquinol, is appreciated as an important lipophilic antioxidant to protect free radical induced damages to DNA, lipid, and proteins. Given that older adults have increased production of free radicals, suboptimal antioxidant defenses toward free radicals, and a decreased capability to replenish utilized CoQ10, CoQ10 supplementation can be one of feasible ways to increase CoQ10 status in order adults. Most supplements available for consumers are in the oxidized form. While the ubiquinol form is also available, whether the reduced form will be more effective to replenish CoQ10 status in older subjects remains to be explored. Thus, investigators aimed to examine whether ubiquinol will be more effectively absorbed in older adults with a low antioxidant defense status. To pursue this aim, investigators will conduct a double blind, randomized, crossover design trail with 5 study visits (1 screening visit and 4 study visits). Ten older men (>55 y, BMI: 25-5 kg/m2) with a compromised antioxidant defenses will be recruited and complete the trial. Eligible subjects will be randomized to receive 200 mg/d ubiquinol or ubiquinone for 2 weeks with 2-week washout between crossover. Ubiquinol and ubiquinone in plasma and immune cells in blood will be assessed to reveal whether the reduced form, ubiquinol, is more absorbable than the oxidized form, ubiquinone in older male adults.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Age: >55 and <76 y
* BMI: ≥25 and <35 kg/m2
* Willing to take the assigned supplement for 4 weeks
* Willing to maintain dietary habit for 6 week
* <1000 µmol/L Fe2+ plasma total antioxidant capacity determined by Ferric Reducing Antioxidant Power and <400 µmol/L total thiol content in plasma

Exclusion Criteria:

* Regular use of any dietary supplements containing vitamins and minerals; however, subjects who are willing to refrain from the use of these supplements for 1 mo prior to their enrollment and throughout the entire study may be considered eligible; subjects will be excluded if they are taking physician prescribed vitamin and/or mineral supplements
* Use of medications known to affect lipid metabolism
* Gain or loss of ≥5% of body weight in the last 6 mo
* Impaired gastrointestinal, renal, and endocrine functions, diseases, conditions or medications influencing gastrointestinal absorption
* Unusual dietary pattern, including vegan/vegetarian
* Active treatment for cancer of any type longer than 1 year.
* Daily alcoholic intake of more than 14 drinks/week (168 oz. beer, 56 oz. wine, 14 oz. hard liquor)
* Values of standard blood biochemistries are critically abnormal based on study physician's

Ages: 56 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-05-17 (Actual)

PRIMARY OUTCOMES:
Concentration change of ubiquinol and ubiquinone in peripheral blood mononuclear cells | before and after the 2-week supplementation of coenzyme Q10
  Concentration change of ubiquinol and ubiquinone in peripheral blood mononuclear cells before and after the 2-week supplementation of coenzyme Q10

SECONDARY OUTCOMES:
Concentration change of ubiquinol and ubiquinone in plasma | before and after the 2-week supplementation of coenzyme Q10
  Concentration change of ubiquinol and ubiquinone in plasma before and after the 2-week supplementation of coenzyme Q10

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Chen, Principal Investigator — Tufts University
Locations (1):
- Oliver Chen, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Y , Liu J , Chen XQ , Oliver Chen CY . Ubiquinol is superior to ubiquinone to enhance Coenzyme Q10 status in older men. Food Funct. 2018 Nov 14;9(11):5653-5659. doi: 10.1039/c8fo00971f. PMID 30302465